CLINICAL TRIAL: NCT04062487
Title: A Clinical Application Study of Mixed Reality Technology Assisted Lumbar Pedicle Screws Implantation
Brief Title: Screws Implantation Assisted With Mixed Reality Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20170109-04
Record Dates: First submitted 2019-08-19; First posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Spine Degeneration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lumbar pedicle screws implantation of traditional procedure (Experimental): traditional method of lumbar pedicle screws implantation
  Interventions: Device: Mixed Reality technology

INTERVENTIONS:
Device: Mixed Reality technology — combine image with real body

SUMMARY:
Prospective comparative study of Mixed Reality Technology（MR）assisted lumbar pedicle screws placement and traditional lumbar pedicle screws placement.

DETAILED DESCRIPTION:
In this study, the randomized controlled method was adopted to prospectively include the samples, and the differences in surgical procedures and efficacy were compared between the thoracolumbar pedicle screw implantation assisted by MR and the traditional thoracolumbar pedicle screw implantation, so as to provide a plan for clinicians to choose the surgical method.

ELIGIBILITY:
Inclusion Criteria:

* Course of disease≥6 months, all patients with lumbago back pain, radiation pain of lower limbs, lumbar disc herniation diagnosed with or without spinal stenosis.
* The course of disease≥6 months, all patients had lumbar back pain, accompanied by or without intermittent claudication, and the diagnosis of lumbar spondylolisthesis was clear, but the vertebral isthmus was not broken.
* The patient's symptoms were consistent with the imaging examination results, failed to respond to conservative treatment, and met the surgical indications.
* The lesion segment is no more than 3 vertebral bodies.
* Preoperative improvement of X-ray, CT, MRI examination.
* Patients without active bleeding and female patients is not in menstrual period.

Exclusion Criteria:

* Lumbar acute infection, lumbar tuberculosis, tumor and other diseases.
* Patients with severe cardiopulmonary insufficiency, intolerance to surgery, diabetes and poor blood glucose control, combined with coagulation dysfunction and other contraindications.
* Vertebral fracture patients.
* Bone Mineral Density (BMD) examination: BMD was measured by dual-energy X- ray absorptiometry at the lumbar spine (L2 ~ L4) and femoral head, and BMD and T values were observed. Abnormal bone mass were excluded according T >- 1 SD

Ages: 38 Years to 53 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2018-10-27 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 6 months
  visual analog scale(0-10 scores) is for pain, 0 represent no pain, 10 score represent the severe pain.
Oswestry Disability Index | 6 months
  Oswestry Disability Index is for movement function, Questionnaire examines
The Standard Of Gertzbein-Robbins | 1 day
  the standard of Gertzbein-Robbins :Ⅰ, self-contained complete within the pedicle nail; Ⅱ, self-contained nail through 2 mm below the cortex; Ⅲ, self-contained nail through 2 mm or greater, cortex < 4 mm; Nail through 4 mm or higher cortex; Ⅳ, self-contained, < 6 mm; Ⅴ, self-contained nail through 6 mm or higher cortex.

CONTACTS AND LOCATIONS:
Locations (1):
- Mixed Reality, Nanjing, Jiangsu, China